CLINICAL TRIAL: NCT02862405
Title: Evaluation of the Perception of Objects and Natural Scenes in People With Vision Loss (Loss of Central or Peripheral Vision)
Brief Title: Perception of Objects and Natural Scenes in People With Vision Loss (ACTIVIS)
Acronym: ACTIVIS
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P009
Record Dates: First submitted 2016-08-02; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Vision Loss
Keywords: Vision loss; Object recognition; Space recognition
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with loss of central vision: Patients coming in ophthalmic consultation will be selected for the study. The diagnosis of this disease is based on clinical examination, and imaging of the retina.Patients with only loss of central vision will be selected.
  Interventions: Other: vision tests
- Patients with loss of peripheral vision: Patients coming in ophthalmic consultation will be selected for the study. Patients with loss of peripheral vision will be selected on the bases of presence of tunnel vision.
  Interventions: Other: vision tests
- Control group: Patients without loss of vision.
  Interventions: Other: vision tests

INTERVENTIONS:
Other: vision tests

SUMMARY:
The loss of central vision causes difficulty not only in reading but also in faces recognition, and in particular in the identification of facial expression, objects or spaces. These visual deficits have been mainly studied in relation with reading, which is the main complaint of these kind of patients. However, there are not enough data regarding perception of objects and spaces in this population. Then, the objectives are to study the visual-spatial abilities in individuals with vision loss, and altered cognitive processes, (2) to develop clinics tools for early detection and quantification of visual-spatial deficits and (3)to understand the capacities of normal peripheral vision in order to test the possibility of potential training for use of peripheral vision when central vision is impaired by an ophthalmic pathology.

ELIGIBILITY:
Inclusion Criteria cases:

* Patients with eye disease causing loss of central or peripheral vision
* French speakers
* Age between 18 and 90 years old
* Written consent
* Health insurance

Inclusion Criteria controls:

* Sex and age matched controls (+/- 5 years)
* French speakers
* Normal visual examination with visual acuity of min 9/10

Exclusion Criteria:

* Psychiatric disease or neurological pathologies
* Communication difficulties (deafness / mutism)
* Drug treatment altering concentration
* Mental deterioration with MMS <24
* Alcoholism or addiction to drugs
* Persons under guardianship

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with eye disease causing loss of central or peripheral vision
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparison of performances in visual tests between different groups according to error rate | at inclusion
  These behavioral studies include a series of short tests of 5 to 10 minutes each (not exceeding 60 minutes with breaks and instructions) in which photos of scenes or isolated objects will be presented in central or peripheral vision using a computer screen or a panoramic screen covering a 180° field.
Comparison of performances in visual tests between different groups according to answer time | at inclusion
  These behavioral studies include a series of short tests of 5 to 10 minutes each (not exceeding 60 minutes with breaks and instructions) in which photos of scenes or isolated objects will be presented in central or peripheral vision using a computer screen or a panoramic screen covering a 180° field.

SECONDARY OUTCOMES:
Estimation of the score of visual acuity by the logMAR chart | at inclusion
Measure of lesion size | at inclusion
Pearson correlation coefficient to determine the correlation between the performance parameters during visual tests (error rate and answer time) and clinical parameters (visual acuity and lesion size) | at inclusion
  These behavioral studies include a series of short tests of 5 to 10 minutes each (not exceeding 60 minutes with breaks and instructions) in which photos of scenes or isolated objects will be presented in central or peripheral vision using a computer screen or a panoramic screen covering a 180° field.

CONTACTS AND LOCATIONS:
Overall Officials: Thi Ha Chau Tran, MD, Principal Investigator — Hospital of the Lille Catholic Institute

IPD SHARING:
Plan to Share IPD: No